CLINICAL TRIAL: NCT00611585
Title: Birmingham Hip Resurfacing System (BHR) Post Approval Study: A Prospective, Multi-Centered Study of the Birmingham Hip Resurfacing System
Brief Title: A Safety and Efficacy Study of the Birmingham Hip Resurfacing System
Acronym: BHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHR
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2024-12

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hip Resurfacing (Other): Birmingham Hip Resurfacing
  Interventions: Device: Birmingham Hip Resurfacing

INTERVENTIONS:
Device: Birmingham Hip Resurfacing — Hip resurfacing system: single use device for hybrid fixation in patients requiring primary hip resurfacing arthroplasty
  Other Names: BHR

SUMMARY:
The purpose of this study is to meet a PMA condition of approval of the BHR System. The study will evaluate the long term safety and effectiveness of the BHR system in patients with non-inflammatory and inflammatory arthritis.

DETAILED DESCRIPTION:
This is a post-approval, prospective, non-randomized, longitudinal, unmasked, multi-center, clinical trial designed to evaluate the longer-term safety and effectiveness of the BHR system. The data collected will permit clinical evaluation for the device performance in improving hip pain, function and range of motion through ten years. The study will permit radiographic evaluation of proper component fixation and alignment maintenance through 10 years post-operative. The incidence of revision is an especially important measure in this study. Data collected will allow analysis of the implant survivorship.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age and skeletally mature
* Patients requiring primary hip resurfacing due to:
* Non-inflammatory arthritis (degenerative joint disease) such as osteoarthritis, traumatic arthritis, avascular necrosis, or dysplasia/DDH
* Inflammatory arthritis such as rheumatoid arthritis
* Subject or his/her legal guardian is willing to consent to participate in the study by signing and dating the approved consent form
* Subject is available for clinical follow-up through at least ten years
* Subject meets none of the exclusion criteria

Exclusion Criteria:

* Subjects with infection or sepsis
* Subjects with any vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or postoperative recovery
* Female subjects of child-bearing age
* Subjects with bone stock inadequate to support the device
* Subjects with known moderate to severe renal insufficiency
* Subjects with known or suspected metal sensitivity (e.g. jewelry)
* Subjects who are immunosuppressed with diseases such as AIDS or persons receiving high doses of corticosteroids
* Subjects with psychological or neurological conditions which would pre-empt their ability or unwillingness to participate in the study
* Subjects who are severely overweight

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-09; Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness evaluation based on incidence of revision, radiographic review and Harris Hip Score | 3 months, 1-10 years

SECONDARY OUTCOMES:
Adverse events | post op through 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Andy Engh, MD, Principal Investigator — Anderson Orthopaedic Clinic; Lawrence Housman, MD, Principal Investigator — Tucson Orthopaedic Institute; John Masonis, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.; Edwin Su, MD, Principal Investigator — Hospital for Special Surgery, New York; John Noble, Jr., MD, Principal Investigator — Center for Orthopaedics; Michael Anderson, MD, Principal Investigator — Aurora Medical Center; Christopher Drinkwater, MD, Principal Investigator — University of Rochester
Locations (7):
- United States (7):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Center for Orthopaedics, Lake Charles, Louisiana
  - Hospital for Special Surgery, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Anderson Orthopaedic Clinic, Alexandria, Virginia
  - Aurora Medical Center, Grafton, Wisconsin